CLINICAL TRIAL: NCT03496090
Title: Randomized Multicentric Controlled Clinical Trial of Parallel Groups to Evaluate the Non-therapeutic Inferiority of a Free Diet With a Progressive Diet, in the Treatment of Non-complicated Acute Diverticulitis
Brief Title: Randomized Multicentric Trial to Evaluate a Free Diet With a Progressive Diet in the Treatment of Acute Diverticulitis (DIVERDIET)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Reina Sofía de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIVERDIET
Record Dates: First submitted 2018-03-27; First posted 2018-04-12 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Diverticulitis; Acute Diverticulitis; Diverticulitis, Colonic; Uncomplicated Diverticular Disease; Diverticulitis of Sigmoid; Diet Modification; Dietary Modification
Keywords: Diverticulitis; Uncomplicated Diverticular Disease; Free diet; Dietary restriction; Acute Diverticulitis
MeSH Terms: conditions — Diverticulitis; Diverticulitis, Colonic | interventions — Diet

STUDY DESIGN:
Intervention Model Description: The study is a randomized, multicentric, controlled with active comparator, parallel group, blind to the evaluator, to demonstrate the non-inferiority in the efficacy and therapeutic and safety of the free diet (group 1) compared to the progressive diet (group 2) in the treatment of uncomplicated acute diverticulitis. This study will be carried out on 134 patients with uncomlpicated acute diverticulitis. The subjects will be randomized in a 1: 1 ratio to receive treatment with progressive diet or diet at free demand. The main analysis will take place two months after the start of treatment.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The patient data will be delivered to the investigator/s of the study of each hospital, who will fill out the Data Collection Notebook (DCN) of each patient and program their controls without information of the group to which the patient has been assigned, as such In this way, the consultations are carried out with blinding of the evaluator (the investigator who will do the controls will not know to which group the patient has been assigned).
  The person in charge of carrying out the statistical analysis will not be able to know to which group the patient has been assigned due to the coding done in the DCN.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free diet (Experimental): Free diet or free demand, being comparable to the normal or zero hospital diet
  Interventions: Other: Free diet
- Progressive diet (Active Comparator): Progressive diet for 7 days, liquid diet for the first three days and soft diet without waste, from the 4th to the 7th day.
  Interventions: Other: Progressive diet

INTERVENTIONS:
Other: Free diet — Free diet or free demand, being comparable to the normal or zero hospital diet
  Other Names: Basal diet
  Arms: Free diet
Other: Progressive diet — Progressive diet for 7 days, liquid diet for the first three days and soft diet without waste, from the 4th to the 7th day.
  Arms: Progressive diet

SUMMARY:
Phase III trial is designed to demonstrate the non-inferiority of a free diet versus a progressive diet in the treatment of acute diverticulitis (AD) without complications. In this study, the effectiveness of the short-term free diet is evaluated, as well as its safety and the quality of life that is perceived in front of the progressive diet.

DETAILED DESCRIPTION:
The study will be carried out in the General Surgery and Gastroenterology Services of the following centers:

* Hospital General Universitario Reina Sofía
* Hospital General Universitario Morales Meseguer de Murcia.
* Hospital Universitario Santa Lucía de Cartagena.
* Hospital General Universitario de Elche.
* Complejo Hospitalario Torrecárdenas de Almería

All patients with increased temperature and acute abdominal pain, as well as clinical suspicion of AD, will be screened for their potential selection in the study. Basic blood tests (hemogram) and abdominal ultrasound will be performed and these guidelines will be followed: if the results indicate complicated AD, it will be excluded from the study; if uncomplicated DA is suspected, blood CRP will be requested; if CRP is less than 5 mg / dl, it will be included in the study and ambulatory treatment will be indicated; if CRP is greater than 5mg / dl, abdominal CT with intravenous contrast will be requested. Result: uncomplicated DA, it will be included in the study and it will be indicated ambulatory treatment or complicated DA, it will be excluded from the study-; those patients with uncomplicated AD, but with risk factors, hospital admission will be recommended, and they may be offered to participate in the study.

If the patient meets the criteria for admission to the study, the attending physician (surgeon on duty) will inform and invite them to participate and after signing the informed consent, their data will be collected and they will be contacted. the person of the hospital, in charge of guarding the list and randomization codes to assign him the corresponding research group: group 1 (free diet) or group 2 (progressive diet) (Annex III), - this group will be delivered of your printed diet and you will be instructed about it, as well as, to all patients, the annotations of pain control and temperature on ad-hoc sheet. The patient data will be delivered to the investigator / s of the study of each hospital, who will fill in the Data Collection Notebook (DCN) of each patient and program their controls without information of the group to which the patient has been assigned, as In this way, the consultations are carried out with blinding of the evaluator (the investigator who will do the controls will not know to which group the patient has been assigned). They will also be asked a quality of life questionnaire SF-12 (baseline) and they will be asked for a blood test with a complete blood count and CRP for the 3rd day of treatment.

Outpatients will be contacted daily by phone during the first 3 days of treatment by the study investigator and between the 3rd and 4th day will go to outpatient surgery for clinical and analytical control (1st consultation), filling in the DCN. The hospitalized patients will follow the same clinical and analytical control by the plant surgeon and the study investigator, filling in the DCN. They will be asked for new blood tests with CRP for the 7th day of treatment and, in those patients who do not have a colonoscopy in the last 12 months prior to entering the study, an endoscopic study will be requested before 60 days for confirmation of diverticular disease, filling in the DCN. They will be given a new SF-12 quality of life questionnaire that they will fill out on the 7th day of the start of the treatment. They will be cited for a new consultation (2nd consultation) to all patients (outpatients and those who have been hospitalized), 30 days of the beginning of the treatment, with new clinical control and annotation of the last analytical, as well as third and last SF-12 quality of life questionnaire, in the DCN. To conclude, patients who were asked for colonoscopy, will be cited in a final consultation (3rd) 2 months after beginning the treatment with the endoscopic result closing the study, with the last entries in the DCN.

Sample size:

To obtain a power of 80% to reject the null hypothesis Ho: that the difference of proportions p1 and p2 is lower than the non-inferiority limit of -10, and taking into account that the level of significance is 5%, assuming that the proportion of non-treatment failure in both treatment groups is 94.7%, the total number of patients expected to be included in the study is 134 patients, with an expected percentage of dropouts of 5%, which 67 patients will receive treatment through free diet and other 67 patients through progressive diet. The endpoint for the main comparison is the proportion of subjects with a lower treatment failure rate at one month (30 days) of follow-up.

Statistical treatment:

The continuous variables will be summarized using descriptive statistics: mean, standard deviation (SD), median, minimum, maximum, number of observations and number of missing observations. Non-normal continuous data will be presented as maximum, top quartile, median, lowest quartile, minimum and number of observations. The categorical variables will be described using absolute and relative frequencies.

For the comparisons between variables, the bivariate analysis will be used. The scores of each dependent variable will be compared with the independent variables using parametric statistical methods (and nonparametric when the parametric application criteria are not met). When the changes within the same treatment group are analyzed, statistical tests for related or paired samples will be used.

In the event that the variables follow the normal distribution, one or more of the following techniques will be described:

- If a variable is of a quantitative type and the other is categorical, for the comparison of the means with a dichotomous variable, the Student's t test will be used. In cases where the qualitative variable has more than 2 categories, the one-way variance analysis (ANOVA) will be used. In the analysis of the variance of a factor with repeated measures, it will be assumed that the subjects are randomly selected from normal populations with the same variance. Previously, the assumptions of independence, normality and equality of variances will be checked.

In the case that the variables do not follow the normal distribution:

* If one variable is quantitative and the other qualitative, the test to be applied will be the Mann-Whitney U test when the qualitative variable has 2 levels, and the Kruskall-Wallis test if the qualitative measurement is formed by 3 levels or plus.
* If both variables are of the categorical type, a cross-tabulation will be performed (contingency tables) using the Pearson chi-square statistic to test the independence hypothesis or the Fisher test (in 2 x 2 tables) ). An analysis of typed residuals corrected will be carried out in order to interpret the meaning of the association detected.

For the non-inferiority analysis in the main variables, a calculation will be made using the Farrington-Manning score, Miettinen-Nurminen Score and Gart-Nam Score tests, with a significance level of 0.05, and a limit of no- inferiority of 0.10. For the continuous variables, non-inferiority will be evaluated by the difference of means with the Mann-Whitney U and the Wilcoxon test.

All statistical comparisons will be made using statistical tests with a level of significance p = 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of uncomplicated acute diverticulitis
* Adequate oral tolerance
* Good response to the first emergency treatment measures (analgesics and antibiotic therapy): improvement of pain and decrease in temperature.
* Willing to continue treatment at home under supervision.
* Accept sign informed consent.

Exclusion Criteria:

* Acute complicated diverticulitis (from grade Ib of the modified Hinchey Classification).
* No good response to the first emergency treatment measures (analgesics and antibiotics): maintenance or increase of abdominal pain, persistence of fever, oral intolerance or vomiting, clinical worsening.
* Antibiotic treatment for diverticulitis in the previous month.
* Suspicion of colorectal cancer.
* Pregnant.
* Refuses to sign informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-04-16 (Actual)

PRIMARY OUTCOMES:
Success in the treatment | 30 days
  Absence of persistence, increase or recurrence of abdominal pain or fever, transition to a stage higher than that of the modified Hinchey classification (requiring radiological drainage and / or surgical treatment), need for hospital admission (for outpatients) and death attributed to this diagnosis.

SECONDARY OUTCOMES:
Pain score | 7 days
  The evaluation in each treatment group of pain intensity, using visual analogue scale (VAS) of pain, self-evaluated daily after dinner. Min value 0. Max value 10. Higher values represent a worse outcome.
Body temperature | 7 days
  Axillary temperature curve, as a reference, by one shot every 12 hours.
PCR value | day 0, 3 and 7
  The comparison in each treatment group of the levels of C-reactive protein (CRP).
Increase in stage | 30 days
  Percentage of patients in each treatment group who pass to a stage higher than Ia in the Hinchey classification modified.
Need for hospital admission | 30 days
  Percentage of outpatients in each treatment group who require hospital admission.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge A Benavides Buleje, Dr., Principal Investigator — Hospital General Universitario Reina Sofía de Murcia
Locations (1):
- Hospital General Universitario Reina Sofía, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tursi A, Elisei W, Brandimarte G, Giorgetti GM, Aiello F. Predictive value of serologic markers of degree of histologic damage in acute uncomplicated colonic diverticulitis. J Clin Gastroenterol. 2010 Nov-Dec;44(10):702-6. doi: 10.1097/MCG.0b013e3181dad979. PMID 20485187
- [Result] Klarenbeek BR, de Korte N, van der Peet DL, Cuesta MA. Review of current classifications for diverticular disease and a translation into clinical practice. Int J Colorectal Dis. 2012 Feb;27(2):207-14. doi: 10.1007/s00384-011-1314-5. Epub 2011 Sep 17. PMID 21928041
- [Result] Biondo S, Golda T, Kreisler E, Espin E, Vallribera F, Oteiza F, Codina-Cazador A, Pujadas M, Flor B. Outpatient versus hospitalization management for uncomplicated diverticulitis: a prospective, multicenter randomized clinical trial (DIVER Trial). Ann Surg. 2014 Jan;259(1):38-44. doi: 10.1097/SLA.0b013e3182965a11. PMID 23732265
- [Result] Reynolds IS, Heaney RM, Khan W, Khan IZ, Waldron R, Barry K. The Utility of Neutrophil to Lymphocyte Ratio as a Predictor of Intervention in Acute Diverticulitis. Dig Surg. 2017;34(3):227-232. doi: 10.1159/000450836. Epub 2016 Dec 10. PMID 27941316
- [Result] Makela JT, Klintrup K, Takala H, Rautio T. The role of C-reactive protein in prediction of the severity of acute diverticulitis in an emergency unit. Scand J Gastroenterol. 2015 May;50(5):536-41. doi: 10.3109/00365521.2014.999350. Epub 2015 Feb 9. PMID 25665622
- [Result] van de Wall BJ, Draaisma WA, van der Kaaij RT, Consten EC, Wiezer MJ, Broeders IA. The value of inflammation markers and body temperature in acute diverticulitis. Colorectal Dis. 2013 May;15(5):621-6. doi: 10.1111/codi.12072. PMID 23088216
- [Result] Nizri E, Spring S, Ben-Yehuda A, Khatib M, Klausner J, Greenberg R. C-reactive protein as a marker of complicated diverticulitis in patients on anti-inflammatory medications. Tech Coloproctol. 2014 Feb;18(2):145-9. doi: 10.1007/s10151-013-1044-5. Epub 2013 Jun 27. PMID 23807310
- [Result] Ferzoco LB, Raptopoulos V, Silen W. Acute diverticulitis. N Engl J Med. 1998 May 21;338(21):1521-6. doi: 10.1056/NEJM199805213382107. No abstract available. PMID 9593792
- [Result] Jackson JD, Hammond T. Systematic review: outpatient management of acute uncomplicated diverticulitis. Int J Colorectal Dis. 2014 Jul;29(7):775-81. doi: 10.1007/s00384-014-1900-4. Epub 2014 May 25. PMID 24859874
- [Result] Martin Gil J, Serralta De Colsa D, Garcia Marin A, Vaquero Rodriguez A, Rey Valcarcel C, Perez Diaz MD, Sanz Sanchez M, Turegano Fuentes F. [Safety and efficiency of ambulatory treatment of acute diverticulitis]. Gastroenterol Hepatol. 2009 Feb;32(2):83-7. doi: 10.1016/j.gastrohep.2008.10.005. Epub 2009 Feb 5. Spanish. PMID 19231679
- [Result] Rosado-Cobian R, Blasco-Segura T, Ferrer-Marquez M, Marin-Ortega H, Perez-Dominguez L, Biondo S, Roig-Vila JV. Complicated diverticular disease: Position statement on outpatient management, Hartmann's procedure, laparoscopic peritoneal lavage and laparoscopic approach. Consensus document of the Spanish Association of Coloproctology and the Coloproctology Section of the Spanish Association of Surgeons. Cir Esp. 2017 Aug-Sep;95(7):369-377. doi: 10.1016/j.ciresp.2017.03.008. Epub 2017 Apr 14. English, Spanish. PMID 28416357
- [Result] Pelaez N, Pera M, Courtier R, Sanchez J, Gil MJ, Pares D, Grandea L. [Applicability, safety and efficacy of an ambulatory treatment protocol in patients with uncomplicated acute diverticulitis]. Cir Esp. 2006 Dec;80(6):369-72. doi: 10.1016/s0009-739x(06)70989-7. Spanish. PMID 17192220
- [Result] Moya P, Arroyo A, Perez-Legaz J, Serrano P, Candela F, Soriano-Irigaray L, Calpena R. Applicability, safety and efficiency of outpatient treatment in uncomplicated diverticulitis. Tech Coloproctol. 2012 Aug;16(4):301-7. doi: 10.1007/s10151-012-0847-0. Epub 2012 Jun 16. PMID 22706731
- [Result] Mizuki A, Nagata H, Tatemichi M, Kaneda S, Tsukada N, Ishii H, Hibi T. The out-patient management of patients with acute mild-to-moderate colonic diverticulitis. Aliment Pharmacol Ther. 2005 Apr 1;21(7):889-97. doi: 10.1111/j.1365-2036.2005.02422.x. PMID 15801924
- [Result] Isacson D, Thorisson A, Andreasson K, Nikberg M, Smedh K, Chabok A. Outpatient, non-antibiotic management in acute uncomplicated diverticulitis: a prospective study. Int J Colorectal Dis. 2015 Sep;30(9):1229-34. doi: 10.1007/s00384-015-2258-y. Epub 2015 May 20. PMID 25989930
- [Result] Etzioni DA, Chiu VY, Cannom RR, Burchette RJ, Haigh PI, Abbas MA. Outpatient treatment of acute diverticulitis: rates and predictors of failure. Dis Colon Rectum. 2010 Jun;53(6):861-5. doi: 10.1007/DCR.0b013e3181cdb243. PMID 20484998
- [Result] van Dijk ST, Rottier SJ, van Geloven AAW, Boermeester MA. Conservative Treatment of Acute Colonic Diverticulitis. Curr Infect Dis Rep. 2017 Sep 23;19(11):44. doi: 10.1007/s11908-017-0600-y. PMID 28942590
- [Result] Vennix S, Morton DG, Hahnloser D, Lange JF, Bemelman WA; Research Committee of the European Society of Coloproctocology. Systematic review of evidence and consensus on diverticulitis: an analysis of national and international guidelines. Colorectal Dis. 2014 Nov;16(11):866-78. doi: 10.1111/codi.12659. PMID 24801825
- [Result] Stollman N, Smalley W, Hirano I; AGA Institute Clinical Guidelines Committee. American Gastroenterological Association Institute Guideline on the Management of Acute Diverticulitis. Gastroenterology. 2015 Dec;149(7):1944-9. doi: 10.1053/j.gastro.2015.10.003. Epub 2015 Oct 8. No abstract available. PMID 26453777
- [Result] Binda GA, Cuomo R, Laghi A, Nascimbeni R, Serventi A, Bellini D, Gervaz P, Annibale B; Italian Society of Colon and Rectal Surgery. Practice parameters for the treatment of colonic diverticular disease: Italian Society of Colon and Rectal Surgery (SICCR) guidelines. Tech Coloproctol. 2015 Oct;19(10):615-26. doi: 10.1007/s10151-015-1370-x. Epub 2015 Sep 16. PMID 26377584
- [Result] Andeweg CS, Mulder IM, Felt-Bersma RJ, Verbon A, van der Wilt GJ, van Goor H, Lange JF, Stoker J, Boermeester MA, Bleichrodt RP; Netherlands Society of Surgery; Working group from Netherlands Societies of Internal Medicine, Gastroenterologists, Radiology, Health echnology Assessment and Dieticians. Guidelines of diagnostics and treatment of acute left-sided colonic diverticulitis. Dig Surg. 2013;30(4-6):278-92. doi: 10.1159/000354035. Epub 2013 Aug 20. PMID 23969324
- [Result] Feingold D, Steele SR, Lee S, Kaiser A, Boushey R, Buie WD, Rafferty JF. Practice parameters for the treatment of sigmoid diverticulitis. Dis Colon Rectum. 2014 Mar;57(3):284-94. doi: 10.1097/DCR.0000000000000075. No abstract available. PMID 24509449
- [Result] Stam MA, Draaisma WA, van de Wall BJ, Bolkenstein HE, Consten EC, Broeders IA. An unrestricted diet for uncomplicated diverticulitis is safe: results of a prospective diverticulitis diet study. Colorectal Dis. 2017 Apr;19(4):372-377. doi: 10.1111/codi.13505. PMID 27611011
- [Result] van de Wall BJ, Draaisma WA, van Iersel JJ, van der Kaaij R, Consten EC, Broeders IA. Dietary restrictions for acute diverticulitis: evidence-based or expert opinion? Int J Colorectal Dis. 2013 Sep;28(9):1287-93. doi: 10.1007/s00384-013-1694-9. Epub 2013 Apr 19. PMID 23604409
- [Result] Andersen JC, Bundgaard L, Elbrond H, Laurberg S, Walker LR, Stovring J; Danish Surgical Society. Danish national guidelines for treatment of diverticular disease. Dan Med J. 2012 May;59(5):C4453. PMID 22549495
- [Result] Sartelli M, Catena F, Ansaloni L, Coccolini F, Griffiths EA, Abu-Zidan FM, Di Saverio S, Ulrych J, Kluger Y, Ben-Ishay O, Moore FA, Ivatury RR, Coimbra R, Peitzman AB, Leppaniemi A, Fraga GP, Maier RV, Chiara O, Kashuk J, Sakakushev B, Weber DG, Latifi R, Biffl W, Bala M, Karamarkovic A, Inaba K, Ordonez CA, Hecker A, Augustin G, Demetrashvili Z, Melo RB, Marwah S, Zachariah SK, Shelat VG, McFarlane M, Rems M, Gomes CA, Faro MP, Junior GA, Negoi I, Cui Y, Sato N, Vereczkei A, Bellanova G, Birindelli A, Di Carlo I, Kok KY, Gachabayov M, Gkiokas G, Bouliaris K, Colak E, Isik A, Rios-Cruz D, Soto R, Moore EE. WSES Guidelines for the management of acute left sided colonic diverticulitis in the emergency setting. World J Emerg Surg. 2016 Jul 29;11:37. doi: 10.1186/s13017-016-0095-0. eCollection 2016. PMID 27478494
- [Result] Kruis W, Germer CT, Leifeld L; German Society for Gastroenterology, Digestive and Metabolic Diseases and The German Society for General and Visceral Surgery. Diverticular disease: guidelines of the german society for gastroenterology, digestive and metabolic diseases and the german society for general and visceral surgery. Digestion. 2014;90(3):190-207. doi: 10.1159/000367625. Epub 2014 Nov 19. PMID 25413249
- [Result] Biondo S, Lopez Borao J, Millan M, Kreisler E, Jaurrieta E. Current status of the treatment of acute colonic diverticulitis: a systematic review. Colorectal Dis. 2012 Jan;14(1):e1-e11. doi: 10.1111/j.1463-1318.2011.02766.x. PMID 21848896
- [Result] Boermeester MA, Humes DJ, Velmahos GC, Soreide K. Contemporary Review of Risk-Stratified Management in Acute Uncomplicated and Complicated Diverticulitis. World J Surg. 2016 Oct;40(10):2537-45. doi: 10.1007/s00268-016-3560-8. PMID 27206400
- [Result] Bugiantella W, Rondelli F, Longaroni M, Mariani E, Sanguinetti A, Avenia N. Left colon acute diverticulitis: an update on diagnosis, treatment and prevention. Int J Surg. 2015 Jan;13:157-164. doi: 10.1016/j.ijsu.2014.12.012. Epub 2014 Dec 11. PMID 25497007
- [Result] Balasubramanian I, Fleming C, Mohan HM, Schmidt K, Haglind E, Winter DC. Out-Patient Management of Mild or Uncomplicated Diverticulitis: A Systematic Review. Dig Surg. 2017;34(2):151-160. doi: 10.1159/000450865. Epub 2016 Oct 5. PMID 27701164
- [Result] Morris AM, Regenbogen SE, Hardiman KM, Hendren S. Sigmoid diverticulitis: a systematic review. JAMA. 2014 Jan 15;311(3):287-97. doi: 10.1001/jama.2013.282025. PMID 24430321
- [Result] Medina-Fernandez FJ, Diaz-Jimenez N, Gallardo-Herrera AB, Gomez-Luque I, Garcilazo-Arsimendi DJ, Gomez-Barbadillo J. New trends in the management of diverticulitis and colonic diverticular disease. Rev Esp Enferm Dig. 2015 Mar;107(3):162-70. PMID 25733040
- [Result] Park HC, Kim BS, Lee BH. Management of right colonic uncomplicated diverticulitis: outpatient versus inpatient management. World J Surg. 2011 May;35(5):1118-22. doi: 10.1007/s00268-011-1048-0. PMID 21409607
- [Result] Diez Buron F, Marcos Vidal JM, Baticon Escudero PM, Montes Armenteros A, Bermejo Lopez JC, Merino Garcia M. [Agreement between verbal numerical scale and visual analog scale assessments in monitoring acute postoperative pain]. Rev Esp Anestesiol Reanim. 2011 May;58(5):279-82. doi: 10.1016/s0034-9356(11)70062-7. Spanish. PMID 21688506
- [Result] Vilagut G, Ferrer M, Rajmil L, Rebollo P, Permanyer-Miralda G, Quintana JM, Santed R, Valderas JM, Ribera A, Domingo-Salvany A, Alonso J. [The Spanish version of the Short Form 36 Health Survey: a decade of experience and new developments]. Gac Sanit. 2005 Mar-Apr;19(2):135-50. doi: 10.1157/13074369. Spanish. PMID 15860162
- [Result] Alonso J, Regidor E, Barrio G, Prieto L, Rodriguez C, de la Fuente L. [Population reference values of the Spanish version of the Health Questionnaire SF-36]. Med Clin (Barc). 1998 Oct 10;111(11):410-6. Spanish. PMID 9834913
- [Result] Schmidt S, Vilagut G, Garin O, Cunillera O, Tresserras R, Brugulat P, Mompart A, Medina A, Ferrer M, Alonso J. [Reference guidelines for the 12-Item Short-Form Health Survey version 2 based on the Catalan general population]. Med Clin (Barc). 2012 Dec 8;139(14):613-25. doi: 10.1016/j.medcli.2011.10.024. Epub 2012 Jan 11. Spanish. PMID 22244683
- [Result] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Result] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Result] Garratt A, Schmidt L, Mackintosh A, Fitzpatrick R. Quality of life measurement: bibliographic study of patient assessed health outcome measures. BMJ. 2002 Jun 15;324(7351):1417. doi: 10.1136/bmj.324.7351.1417. PMID 12065262
- See also: hospital diets — https://www.universidadviu.es/dietas-hospitalarias/
- See also: Diverticular Disease: An Update on Pathogenesis and Management. Gut Liver — http://www.gutnliver.org/journal/view.html?doi=10.5009/gnl16552